CLINICAL TRIAL: NCT06334211
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single-center, Single and Multiple Ascending Oral Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of FP-020 in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics, of Single and Multiple Ascending Doses of FP-020 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Collaborators: InClin, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FP-020C-23-001
Record Dates: First submitted 2024-03-01; First posted 2024-03-27 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Phase I; Safety and Tolerability; Pharmacokinetics; Randomized; Single & Multiple Ascending Oral Dose; Placebo-Controlled; Double Blinded; FP-020

STUDY DESIGN:
Intervention Model Description: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single-center, Single and Multiple Ascending Oral Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of FP-020 in Healthy Volunteers
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind (placebo appears the same as active FP-020)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FP-020 (Experimental): 100 mg capsule
  Interventions: Drug: FP-020
- placebo (Placebo Comparator): placebo capsule
  Interventions: Other: placebo

INTERVENTIONS:
Drug: FP-020 — MMP-12 inhibitor
  Arms: FP-020
Other: placebo — placebo
  Arms: placebo

SUMMARY:
This is a study to Investigate the Safety, Tolerability, and Pharmacokinetics, of Single (including Food Effect) and Multiple Ascending Doses of FP-020 in Healthy Adult Volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, first-in-human (FIH), 2-part (Part 1 and Part 2), single-center, randomized, double-blind, placebo-controlled, single ascending dose (SAD)/multiple ascending dose (MAD) study designed to evaluate the safety, tolerability, PK, and food effect of FP-020 in healthy male and female subjects.

Up to 72 healthy male and female adults, including 40 subjects in Part 1 (SAD) and 32 in Part 2 (MAD) will be randomized. Part 1 will include up to 5 SAD cohorts comprised of 8 subjects each, inclusive of 1 food effect (FE) cohort. Part 2 will include up to 4 MAD cohorts comprised of 8 subjects each.

Part 1 - Single Ascending Dose:

Following the Screening Period (Day -28 to Day 2), eligible subjects will be admitted to the CRU on Day 1 to confirm eligibility and to begin an overnight fast before the start of study procedures on Day 1.

Eligible subjects will be randomized to treatment within 1 of 5 sequentially ascending dose cohorts within 24 hours before the administration of study drug on Day 1.

Dose Ascending Cohorts 1a to 1d:

Within each cohort, subjects will be assigned to receive a single dose of FP 020 or placebo on Day 1 in a 6:2 randomization ratio (i.e., 6 to FP-020 and 2 to placebo).

Sentinel dosing will occur within each cohort, whereby on Day 1, the first 2 subjects will receive FP-020 or placebo as assigned per the 1:1 randomization schedule. Following review by the Principal Investigator (PI) or suitably qualified sub-investigator of all available safety data obtained from these 2 sentinel subjects over the first 24 hours post dose, the remaining 6 subjects in each ascending dose cohort will be randomly assigned to receive FP-020 or placebo in a 5:1 ratio on Day 3 in the morning.

Subjects will receive their assigned dose on Day 1 under fasting conditions (10 hours) and complete postdosing procedures as detailed in the Schedule of Assessments. Subjects will remain in the unit for 72 hours (i.e., until Day 4) and will return to the clinic on Day 8 (± 2 days)/End of Study (EOS) or Early Termination (ET) visit for follow-up safety assessments.

Food Effect Cohort 1e:

The FE Cohort will be initiated when SAD Cohorts 1a to 1d have been completed and will be dosed at one of the doses used in one of these cohorts. Sentinel dosing will therefore not be required, as safety and tolerability at this dose will have already been established.

For the FE Cohort 1e, subjects will remain in the CRU from Day -1 through Day 11. Subjects will be randomized (on Day 1 or Day 1) to receive their assigned study drug (FP-020 or placebo) at the same dose in a cross-over fashion (once fasted [Treatment Period 1] and once fed [Treatment Period 2]) on Day 1 and Day 8, respectively. The 2 periods will be separated by at least 6 days.

Administration of study drug under fed conditions will entail dosing 30 minutes after commencing a standard high-calorie breakfast (subjects are to consume the high-calorie meal within 30 minutes entirely).

Subjects will remain in the unit until Day 11 and will return to the clinic on Day 15 (± 2 days)/EOS visit for follow-up safety assessments.

Part 2 - Multiple Ascending Dose:

Part 2 may be initiated after at least 2 Part 1 SAD cohorts have completed dosing, at a dose determined by the SMC based on safety and PK data from these SAD cohorts.

Following the Screening Period (Day -28 to Day 2), eligible subjects will be admitted to the CRU on Day -1 to confirm eligibility.

On Day 1 or Day 1, eligible subjects will be randomized to treatment into 1 of the sequential cohorts in Part 2.

Within each cohort, subjects will be randomized to receive once daily dose of FP-020 or placebo in a 6:2 ratio in the CRU for 10 days. Subjects will receive their assigned treatment in the morning under fasting conditions.

Sentinel dosing will occur within each cohort, whereby on Day 1, the first 2 subjects will be assigned to receive FP-020 or placebo in a 1:1 randomization ratio. Following PI review of the safety data obtained in these 2 "sentinel" subjects over the first 48 hours, the remaining 6 subjects in each cohort will be randomly assigned to receive FP-020 or placebo for 10 days in a 5:1 ratio starting on Day 4 in the morning.

Subjects in Part 2 will be confined in the CRU from Days -1 to 13. Subjects will return to the CRU on Day 17 (± 2 days)/EOS visit for follow-up safety assessments.

The recommended dose for each MAD cohort and the final number of Part 2 MAD cohorts will be determined by the Safety Monitoring Committee (SMC) following the blinded review of the available PK and safety data from Part 1 and preceding cohort(s) in Part 2. The decision to proceed to each successive dose level will be based on blinded assessment of all available safety and PK data by the SMC. Each follow-on cohort will not commence dosing until a minimum of 7 subjects from the prior cohort have completed their in-house/confinement period. Also, dosing of the next cohort will not occur until at least 7 days have elapsed since dosing of the previous cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 years and ≤ 60 years of age at the time of signing informed consent.
2. Subjects must be in good general health in the opinion of the Investigator, with no significant medical history, no clinically significant abnormalities on physical examination, vital signs, ECG, and laboratory safety tests performed at Screening and/or before administration of the first dose of study drug.
3. Clinical laboratory test values within normal ranges or < 1.5 times the upper limit of normal (ULN) as specified by the testing laboratory unless deemed not clinically significant (NCS) by the Investigator, with the exception of bilirubin as described below.
4. Nonsmoker or ex-smoker who has discontinued smoking and/or use of nicotine containing products for at least 6 months prior to the first dose of study drug, confirmed by a negative cotinine test at Screening and Day -1. Note however that casual smoking (e.g., 5 cigarettes [or equivalent] per week) is permitted during that period (i.e., within 3 months prior to dosing) as long as the cotinine test on Day 1 is negative.
5. Ability to communicate well with the Investigator, in the local language, and to understand and comply with the requirements of the study.
6. Body mass index (BMI) within the range 18 to 32 kg/m2 (inclusive).
7. Females of childbearing potential and not abstinent must be willing to use a double barrier contraceptive method (progesterone-only hormone contraceptive [oral, injectable, implantable], intrauterine device [IUD], diaphragm, cervical cap, contraceptive sponge, condom) and refrain from oocyte donation from screening to 30 days after the last dose of study intervention. Estrogen-containing products are not allowed. Females who are abstinent are not required to use a contraceptive method unless they become sexually active. Alternatively, females must be postmenopausal for ≥1 year or surgically sterile (with tubal ligation, hysterectomy, or bilateral oophorectomy) for ≥6 months, confirmed by FSH level >40mIU at Screening. Note that females on HRT are not eligible.
8. Males with female partners of childbearing potential will agree to use barrier contraceptive (i.e., condom) and their female partners must use a highly effective method of contraception from screening to 90 days after the last dose of study drug. Males must also refrain from sperm donations during this time period. Males who are abstinent will not be required to use a contraceptive method unless they become sexually active.
9. Subjects capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

1. Recent (less than 6 weeks) wound, or presence of an ongoing non-healing skin wound.
2. Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would significantly alter the absorption, metabolism, or elimination of drugs; constitute a risk when taking the study intervention; interfere with the interpretation of data; or would make it unlikely that the subject will complete the study per protocol.
3. Active malignancy and/or history of malignancy in the past 5 years, with the exception of completely excised non-melanoma skin cancer or low grade cervical intraepithelial neoplasia.
4. Serious local or systemic infection within 1 month of Screening requiring antibiotic treatment or history of recurrent infections.
5. Surgery within the past 3 months prior to the first dose of study drug administration determined by the Investigator to be clinically relevant.
6. The subject has a history of severe drug allergy or hypersensitivity or food allergy, including anaphylaxis.
7. The subject has donated more than 1 unit (500 mL) of blood within 4 weeks prior to the first dose of study drug.
8. Positive for human immunodeficiency virus (HIV) antibody or antigen.
9. Positive hepatitis C virus (HCV) antibody or positive hepatitis B surface antigen (HBsAg).
10. Positive urine drug screen/alcohol breath test on Day -1 (admission). Repeat urine drug screens will be permitted for suspected false positive results.
11. Positive COVID-19 test (conducted as per institutional guidelines).
12. Abnormal vital signs (resting heart rate < 40 or > 100 bpm; resting systolic blood pressure >150 or < 90 mmHg or diastolic blood pressure > 90 or < 50 mmHg) at Screening or before administration of the first dose of study drug.
13. Any other abnormal vital signs that are considered to be clinically significant by the Investigator.
14. QTcF interval (QT with Fridericia's correction) > 450 msec in males and > 470 msec in females (based on the mean of triplicate measurements taken at screening), cardiac arrhythmia, or any clinically significant abnormality in the resting ECG as deemed by the Investigator.
15. Females with heavy menstruating cycles and borderline-low iron studies.
16. Alanine transaminase (ALT) or aspartate aminotransferase (AST) >1.5 upper limit of normal.
17. Bilirubin outside of the normal range (total bilirubin between 0.1 and 1.2 mg/dL (1.71 to 20.5 µmol/L).
18. Creatinine clearance < 90 mL/min (estimated from Cockcroft Gault equation).
19. Subject is pregnant, lactating, or is planning to become pregnant during the study.
20. Inability to tolerate oral medications.
21. All prescription and over-the-counter medications (including herbal medications) except for non-estrogen contraceptives, are prohibited within 7 days before dosing through EOS.
22. Any estrogen-containing products, e.g., contraceptives, patches, creams, implants, within 14 days prior to administration of the first dose of study drug through EOS.
23. Live vaccine(s) within 1 month before Screening or plans to receive such vaccines during the study.
24. Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) before dosing.
25. Current participation in any other investigational drug study or receipt of an investigational drug within 30 days or 5 half-lives (whichever is longer) before dosing.
26. Significant weight loss or gain between Screening and administration of first dose of study drug.
27. Blood donation or significant blood loss within 60 days prior to administration of first dose of study drug.
28. Plasma donation within 7 days prior to administration of first dose of study drug.
29. Diets that could alter metabolism (i.e., high protein, Slim Fast®, Nutrisystem®, etc.) within 7 days prior to administration of first dose of study drug.
30. History or presence of alcohol or drug abuse (including recreational marijuana use) within 1 year prior to administration of first dose of study drug and unwillingness to abstain during the dosing period.
31. Intake of alcohol or caffeine-containing products 48 hours before administration of first dose of study drug.
32. Use of tobacco products (e.g., cigarettes, e-cigarettes, cigars, smokeless tobacco) confirmed by a positive cotinine test on Day -1.
33. Failure to satisfy the Investigator of fitness to participate for any other reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
The incidence, severity, and type of Adverse Events (AEs) and Serious Adverse Events (SAEs). | Part 1 - up to 10 days and Part 2 - up to 17 days
  * Treatment-emergent AEs up to End of Study (EOS)
  * Treatment-emergent AEs leading to premature discontinuation of study drug
  * Treatment-emergent SAEs up to EOS
  * Incidence of DLTs per dose level
Clinically significant abnormalities. | Part 1 - up to 10 days and Part 2 - up to 17 days
  Clinically significant abnormalities in physical examination, vital signs, 12-lead Electrocardiograms (ECGs), and safety laboratory results.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of FP-020 after single, ascending oral doses - Cmax | Single ascending dose (Part 1) - up to 10 days
  Cmax (Maximum concentration)
Pharmacokinetic (PK) profile of FP-020 after single, ascending oral doses - Tmax | Single ascending dose (Part 1) - up to 10 days
  Tmax (Time to maximum concentration)
Pharmacokinetic (PK) profile of FP-020 after single, ascending oral doses - AUC0-24 hours | Single ascending dose (Part 1) - up to 1 day
  AUC0-24 (Area under the curve time 0 to 24 hours)
Pharmacokinetic (PK) profile of FP-020 after single, ascending oral doses - AUC0 - last | Single ascending dose (Part 1) - up to 10 days
  AUC0-last (Area under the curve - to last time collected)
Pharmacokinetic (PK) profile of FP-020 after single, ascending oral doses - AUC0-inf | Single ascending dose (Part 1) - up to 10 days
  AUC0-inf (Area under the curve - extrapolated to infinity)
Pharmacokinetic (PK) profile of FP-020 after single, ascending oral doses - λz | Single ascending dose (Part 1) - up to 10 days
  λz (terminal elimination rate constant)
Pharmacokinetic (PK) profile of FP-020 after single, ascending oral doses - t1/2 | Single ascending dose (Part 1) - up to 10 days
  t1/2 (half-life)
Evaluate the food effect on the PK profile of FP-020 - Cmax | Single ascending dose (Part 1) - up to 10 days
  Cmax in fed vs fasted state
Evaluate the food effect on the PK profile of FP-020 - Tmax | Single ascending dose (Part 1) - up to 10 days
  Tmax in fed vs fasted state
Evaluate the food effect on the PK profile of FP-020 - AUC | Single ascending dose (Part 1) - up to 10 days
  AUC in fed vs fasted state
Evaluate the PK profile of FP-020 after multiple ascending oral doses in healthy subjects - Cmax | Multiple ascending dose (Part 2) - up to 10 days
  Cmax on Day 1 and Day 10
Evaluate the PK profile of FP-020 after multiple ascending oral doses in healthy subjects - Tmax | Multiple ascending dose (Part 2) - up to 10 days
  Tmax on Day 1 and Day 10
Evaluate the PK profile of FP-020 after multiple ascending oral doses in healthy subjects - AUC0 - 24 | Multiple ascending dose (Part 2) - up to 10 days
  AUC0-24 on Day 1 and Day 10
Evaluate the PK profile of FP-020 after multiple ascending oral doses in healthy subjects - AUCo - last | Multiple ascending dose (Part 2) - up to 10 days
  AUC0-last on Day 1 and Day 10
Evaluate the PK profile of FP-020 after multiple ascending oral doses in healthy subjects - AUC0 - inf | Multiple ascending dose (Part 2) - up to 10 days
  AUC0-inf on Day 1 and Day 10
Evaluate the PK profile of FP-020 after multiple ascending oral doses in healthy subjects λz | Multiple ascending dose (Part 2) - up to 10 days
  λz on Day 10
Evaluate the PK profile of FP-020 after multiple ascending oral doses in healthy subjects - t1/2 | Multiple ascending dose (Part 2) - up to 10 days
  t1/2 on Day 10
Evaluate the PK profile of FP-020 after multiple ascending oral doses in healthy subjects - RCmax | Multiple ascending dose (Part 2) - up to 10 days
  RCmax (ratio of Day 10 and Day 1 Cmax values)
Evaluate the PK profile of FP-020 after multiple ascending oral doses in healthy subjects - RAUC | Multiple ascending dose (Part 2) - up to 10 days
  RAUC (ratio of Day 10 and Day 1 AUC0-24 values)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Whitaker, BSN, Study Director — Senior Director of Clinical Operations
Locations (1):
- Scientia Clinical Research Ltd, Randwick, New South Wales, Australia